CLINICAL TRIAL: NCT00914914
Title: A Phase I Trial of p28 (Cell Penetrating Peptide) in the Treatment of Refractory Solid Tumors
Brief Title: Safety Study of a Cell Penetrating Peptide (p28) to Treat Solid Tumors That Resist Standard Methods of Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Tapas K. Das Gupta (Industry)
Responsible Party: Sponsor-Investigator, Dr. Tapas K. Das Gupta, Co-founder, CDG Therapeutics, Inc.
Organization: CDG Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDGTI-p28-001; IND 77754 (Registry Identifier: FDA); 2008-0213 (Other: University of Illinois at Chicago COM IRB); PAF 2009-03370 (Other: University of Illinois at Chicago ORS)
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Refractory Solid Tumors
MeSH Terms: interventions — Interleukin-27; Azurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- p28 Phase I Safety (Experimental): A total of 15 patients were administered p28 i.v. as a short infusion three times per week for 4 weeks followed by a 2-week rest under an accelerated titration 3þ3 dose escalation design.
  Interventions: Drug: p28

INTERVENTIONS:
Drug: p28 — p28 will be dissolved in normal saline and infused intravenously into the patient over 15-30 minutes.
  Other Names: azurin

SUMMARY:
The purpose of this study is to evaluate the safety of an experimental drug (p28) as a treatment for certain advanced cancers which express a protein called p53 and which have not responded to prior treatment.

DETAILED DESCRIPTION:
The drug used in this study is p28, a cancer cell killing peptide. A peptide is a compound made of amino acids, which are substances that the body uses to make protein. The p28 peptide was created from a protein called azurin. Azurin is created by a common disease-causing bacteria named Pseudomonas Aeruginosa. p28 is experimental and has not yet been tested in humans and has not been approved by the FDA for use in cancer subjects.

Up to 30 subjects may be enrolled in order to find 15 subjects who qualify for the study.

Subjects will be enrolled in groups of three, each starting at one of five progressively higher dosage groups. The first group of three subjects will receive the lowest dose of p28 three times a week injected into a vein for four weeks. They will then be monitored for two weeks. If no bad side effects are recorded, the initial three subjects will then receive the second (higher) dose level of p28 three times a week for another four weeks, followed, again, by two weeks of follow up. Additionally, three new subjects will be added to the study and receive p28 on the same schedule, although this second group will start with the second dose level. In this manner, 3 new subjects will be added every six weeks and start treatment at the dose level to which previously enrolled groups have now progressed.

Subjects will be monitored weekly during their first six weeks and then every two weeks for the remainder of the study. Monitoring will include physical exams, blood tests, EKG, and appropriate radiographic imaging (CT, MRI, PET scan, and/or chest X-ray).

The entire study should take 32 weeks for subjects starting at dose 1, 26 weeks for subjects starting at dose 2, 20 weeks for subjects starting at dose 3, 14 weeks for subjects starting at dose 4, and 8 weeks for subjects starting at dose 5 (there is an additional 2 week follow-up period at the end of the study for all subjects included in these figures). All surviving subjects however, will be followed according to the normal follow-up schedule for such subjects at the UIC Oncology Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven solid tumor disease with documentation of measurable metastatic disease as defined by RECIST.
* The term refractory solid tumor signifies patients with metastatic solid tumors who have failed all standard therapy or for whom no standard therapy exists.
* In patients with refractory solid tumors, a pretreatment biopsy (either of the original primary or metastatic deposit) must show p53 (wild-type and to an extent mutant) expression by means of immunocytochemistry.
* Patients must have distant metastases or unresectable local disease, but a projected life expectancy of at least 6 months.
* Patients must have signed an informed consent.
* This study is confined to adults of both sexes, age 18 or older.
* Patients must have no medical problems that would pose an undue risk or that would limit full compliance with the study.
* A minimum of 4 weeks must have elapsed since the completion of prior therapy, including hormonal therapy, chemotherapy, radiation therapy, immunotherapy, oral tyrosine kinase inhibitors and monoclonal antibodies.
* Adequate baseline organ function assessed by the following laboratory values within 30 days prior to study entry:

  * Granulocyte count >1,500/mm3, hematocrit >30%, and platelets >100,000/mm3.
  * Calculated creatinine clearance >50ml/min.
  * Adequate liver function with SGOT, SGPT, LDH, and alkaline phosphatase <3 x the upper limit of normal; serum bilirubin <2.0 mg/dl.
  * PT and PTT not more than 1.5 times the upper limit of normal.
* Adequate cardiac and pulmonary function. Patients with decreased LVEF or PFTs will be evaluated by a cardiologist or pulmonary physician prior to enrollment of this protocol.

Exclusion Criteria:

* Patients who are undergoing chemotherapy or immunotherapy, i.e., cytokines
* Patients with refractory solid tumors whose primary tumor or metastatic deposits do not express p53 (null) will not be eligible.
* Patients with serious additional illness, including HIV, hepatitis, or untreated active infection.
* Patients with any underlying conditions that would contraindicate therapy with the study agent.
* Patients with a history of prior malignancy in the past five years other than the current problem for which he/she is being considered for this trial (patients with prior history of basal cell carcinoma or squamous cell skin cancer are eligible).
* Patients with any other serious medical, i.e., cardiovascular, uncontrolled diabetes (insulin resistant), or psychiatric illness that would prevent informed consent will not be eligible to participate in the study.
* Patients who are either pregnant or lactating (all patients of childbearing potential will receive a pregnancy test within 2 days of study initiation).
* Brain Metastases, current or past (unless treated at least one year prior to enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Clinical and laboratory adverse reactions will be closely monitored by periodic physical and laboratory examination. | 32 weeks
Grade 3 non-hematologic or Grade 4 hematologic toxicity will also define the Maximum Feasible Dose (MFD). | 32 weeks

SECONDARY OUTCOMES:
Reduction in the size of measurable tumors using the RECIST criteria and, if possible, demonstration of p28 localization and biopsy of tumor. | 32 weeks
Calculate peak (serum) concentration of p28 and compare with any sign of toxicity and response. | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Warso, M.D., Principal Investigator — University of Illinois Department of Surgical Oncology
Locations (1):
- University of Illinois at Chicago Department of Surgical Oncology, Chicago, Illinois, United States

REFERENCES:
- [Background] Warso MA, Richards JM, Mehta D, Christov K, Schaeffer C, Rae Bressler L, Yamada T, Majumdar D, Kennedy SA, Beattie CW, Das Gupta TK. A first-in-class, first-in-human, phase I trial of p28, a non-HDM2-mediated peptide inhibitor of p53 ubiquitination in patients with advanced solid tumours. Br J Cancer. 2013 Mar 19;108(5):1061-70. doi: 10.1038/bjc.2013.74. Epub 2013 Feb 28. PMID 23449360